CLINICAL TRIAL: NCT06078332
Title: Reliability of Remote Neuropsychological Assessment in People With Cognitive Disorders
Brief Title: Remote Cognitive Multidomain Assessment in People With Cognitive Disorders
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Chiara Zucchella, Psychologist, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: NPSTV
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Dementia; Cognitive Disorders; Neuropsychological Tests; Cognitive Assessment
Keywords: Remote neuropsychological assessment; Telemedicine; Cognitive impairment; Dementia; Domain-specific neuropsychological tests
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Remote assessment first: Participants will perform the first neuropsychological assessment remotely via video conferencing. After 15 days, the participants will repeat the same neuropsychological tests (second assessment) face to face. Finally, participants and caregivers will complete online the satisfaction questionnaire about remote administration.
- Face-to-face assessment first: Participants will perform the first neuropsychological assessment in presence in the hospital. After 15 days, the participants will repeat the same neuropsychological tests (second assessment) remotely via video conferencing. Finally, participants and caregivers will complete online the satisfaction questionnaire about remote administration .

SUMMARY:
Digital medicine is a useful clinical resource for people with cognitive disorders. Scientific literature has shown that in people with dementia neuropsychological instruments administered in remote are characterized by high psychometric quality and satisfaction levels. However, evidence about the reliability of remote neuropsychological domain-specific tests is still limited in the Italian context.

The principal aims of the study will be 1) to evaluate the reliability of the remote administration of neuropsychological screening and domain-specific tests compared to the face-to-face administration in patients with cognitive disorders; 2) to assess the feasibility and level of satisfaction of patients and caregivers about remote administration.

All participants will be submitted to both face-to-face and remote neuropsychological assessment (by videoconference) in a counterbalanced cross-over design. Finally, all patients and/or caregivers will complete a satisfaction questionnaire about the remote administration.

DETAILED DESCRIPTION:
The pilot study will enroll consecutive patients referring to the Center for cognitive disorders and dementia, UOC Neurology A of the AOUI Verona. For all participants will be obtained a written informed consent after a detailed information during the visit of normal clinical practice.

All patients included will be submitted (in presence or remotely) to a screening assessment of global cognition and level of autonomy in daily life. People with subjective or milder cognitive disorders will be also submitted to a standardized battery of neuropsychological tests aimed at the investigation of specific cognitive areas (memory, attention, executive functions, etc.) (T0). After 15 days (T1) each participant will repeat the same assessment in the mode of administration opposite to the previous one. So, all participants will be submitted to both face-to-face and remote neuropsychological assessment in a counterbalanced cross-over design to reduce the learning bias; half of the participants will perform the first assessment in presence, the other half the first assessment in remote mode. The two neuropsychological assessments will be administered by two psychologists independently.

Finally, all patients and/or caregivers completed a satisfaction questionnaire about the remote administration.

Presence assessment will be carried out in the hospital clinic, according to the normal procedures of good clinical practice. Remote assessment will be carried out through the Virtual Care - Pohema telemedicine platform (developed by GPI SpA), using its function of televisit. The selected neuropsychological instruments are paper-and-pencil and oral tests; the material will be presented to participants via screen sharing.

To assess the reliability of the neuropsychological tests administered in remote mode, the quantitative scores corrected by age, education, and sex (normative tables) will be considered and the statistical analysis Paired Sample T-Test will be used. Graphic comparisons will also be made using the method described by Bland and Altman and Intraclass Correlation Coefficients (ICC) will be calculated.

To assess the feasibility and satisfaction level of patients and caregivers related to remote administration, will be calculate the absolute and relative frequencies of the 2 modes of response (disagreement, agreement) to the 14 questions of the questionnaire developed ad hoc.

ELIGIBILITY:
Inclusion Criteria:

* Being in care at the CDCD of the Verona hospital;
* Diagnosis of Major Neurocognitive Disorder, Mild Neurocognitive Disorder, or Subjective Cognitive Disorder according to DSM 5 criteria;
* Availability of a caregiver for technical support;
* Availability of a device equipped with camera and microphone and internet connection to do the video call;
* Informed consent signed by the patient, the legal representative if present, and the caregiver.

Exclusion Criteria:

* Severe sensory deficits;
* Non-native Italian speakers;
* Primary Psychiatric Disorder;
* MMSE score less than 10;
* Severe Behaviour and Psychological Symptoms of Dementia that limit collaboration;
* Aphasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll consecutive patients referring to the Center for cognitive disorders and dementia of the Verona Hospital (AOUI Verona, Neurology A), already diagnosed with Major Neurocognitive Disorder, Mild Neurocognitive Disorder, or Subjective Cognitive Disorder according to the DSM 5 diagnostic criteria (APA, 2013), regardless of the etiological diagnosis of disease.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Comparison of the remote and face-to-face performance on the Mini-Mental State Examination (MMSE) | Day 1 (t0) and Day 15 (t1)
  The MMSE is a screening test of global cognition that includes tasks designated to asses space-temporal orientation, concentration, attention, verbal memory, naming and visuospatial skills. MMSE is scored from 0 to 30. The cut-off is 24 points. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-24 points) cognitive impairment (Folstein et al., 1975; Magni et al., 1996).
  In the remote assessment the visual stimuli (tasks of reading and copy of drawing) will be displayed on the video using the share screen option.
Comparison of the remote and face-to-face performance on the Activities of Daily Living (ADL) scale | Day 1 (t0) and Day 15 (t1)
  The ADL scale is an informant-based instrument that assesses the level of independence in six basic self-care functions: bathing, dressing, going to toilet, transferring, feeding, and continence. The total score ranges from 0 to 6; one point is given for each skill retained (0=complete dependence, 6=complete independence). The questionnaire can be completed by the patient or the caregiver (Katz et al., 1963).
Comparison of the remote and face-to-face performance on the Instrumental Activities of Daily Living (IADL) scale | Day 1 (t0) and Day 15 (t1)
  The IADL scale was developed to assess the person's level of independence in more complex activities (termed "instrumental activities") necessary for functioning in community settings. The graded scale measures 8 domains of function: telephone use, shopping, cooking, food preparation, housekeeping, laundering, taking drugs, and managing finances. Historically, women were scored on all 8 areas of function; men were scored in only 5 domains. One point is given for each skill retained. The total score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men. The questionnaire can be completed by the patient or the caregiver (Lawton e Brody, 1969).
Comparison of the remote and face-to-face performance on the Rey Auditory Verbal Learning Test (RAVLT) | Day 1 (t0) and Day 15 (t1)
  The RAVLT evaluates verbal learning and memory. The test is designed as a list-learning paradigm and includes three tasks: 1) "immediate recall" (score range from 0-75); 2) "delayed recall" (score range from 0-15); 3) "recognition". The score is given by the number of words correctly remembered; higher the score, better the performance. Omissions and false positives are also counted in the recognition task (Carlesimo et al., 1996).
Comparison of the remote and face-to-face performance on the Forward and Backward Digit Span (DS) test | Day 1 (t0) and Day 15 (t1)
  The Forward and Backward DS tasks are used to assess verbal short-term memory and working memory respectively. The DS tests requires that participants listen to a series of digits and repeat the series in correct forward or backward order. The score is the length of the longest correctly repeated sequence. Higher the score, better the performance (Monaco et al., 2015).
Comparison of the remote and face-to-face performance on the Clock Drawing Test (CDT) | Day 1 (t0) and Day 15 (t1)
  The CDT is used to quickly assess visuospatial, praxis, mental representation, planning and logical abilities. The person is asked to put the numbers on the watch, and then draw the hands to indicate a given moment. The maximum possible score is 10 points. The cut-off point is determined by the age and years of schooling of the person; higher scores indicate better performance (Mondini et al., 2003).
  In the remote assessment the participant will draw the clock on a blank sheet and then show it to the camera.
Comparison of the remote and face-to-face performance on the Frontal Assessment Battery (FAB) | Day 1 (t0) and Day 15 (t1)
  The FAB is a short tool for the assessment of executive functions consisting of six subtests that explore different abilities related to the frontal lobes (Similarities, Lexical Fluency, Motor Series, Conflicting Instructions, Go-No-Go, Prehension Behaviour). The sum of the sub-scores from each of the six components are added up to generate total score out of 18. Higher scores indicate better performance; the cut-off point is 12 (Aiello et al., 2021).
Comparison of the remote and face-to-face performance on the Stroop Color and Word Test (SCWT) | Day 1 (t0) and Day 15 (t1)
  The SCWT assesses selective attention and the ability to inhibit cognitive interference. People examined are required to read three different tables as quickly as possible. Two of them represent the congruous conditions (word reading, color naming), the third table represent the interference condition (named color-word). The two total scores "interference time" and "interference errors" are calculated from the completion times and number of errors for each condition by a formula. Higher scores indicate worst performance (Caffarra et al., 2002).
  In the remote assessment the stimuli will be displayed on the video using the share screen option.
Comparison of the remote and face-to-face performance on the Raven's Coloured Progressive Matrices (CPM) test | Day 1 (t0) and Day 15 (t1)
  The Raven's CPM is a culture-fair test of nonverbal intelligence. The test includes 36 items that are divided into three sets of 12 (set A, Ab and B), in order of increasing difficulty within each set. The person is shown a large square that contains a pattern with a piece missing and is asked to complete the pattern by choosing the correct option from six available pieces. The score corresponds to the total number of matrices that have been successfully completed. Higher scores indicate better performance (Basso et al., 1987).
  In the remote assessment the visual stimuli will be displayed on the video using the share screen option.
Comparison of the remote and face-to-face performance on the Phonemic Verbal Fluency test | Day 1 (t0) and Day 15 (t1)
  The Phonemic Verbal Fluency test assess the phonological lexical access performance. In the task examinees are asked to orally produce as many words beginning with a given letter (F, A and S) as possible in sixty seconds. The total score is obtained from the sum of the number of valid words produced for each letter. Higher scores indicate better performance (Carlesimo et al., 1996).
Comparison of the remote and face-to-face performance on the Semantic Verbal Fluency test | Day 1 (t0) and Day 15 (t1)
  The Semantic Verbal Fluency test assess the semantic lexical access performance. In the task examinees are asked to orally produce as many words from a specific category (animals, fruit, vehicles) as possible in sixty seconds. The total score is obtained from the sum of the number of valid words produced for each category. Higher scores indicate better performance (Novelli et al., 1986).
Comparison of the remote and face-to-face performance on the Constructional Praxis test | Day 1 (t0) and Day 15 (t1)
  The Constructional Praxis test assess visuoconstructive abilities. In particular, the ability to copy geometric forms, as well as visual planning skills. The test is composed of seven images of different geometric figures that are progressively more complex in terms of their shape. The examinees is asked to copy each figure once at a time, in the most accurate way possible. A drawing is considered correct (and receives 2 points) when the overall shape is reproduced. Each incorrect drawing receives the score of 1 or 0 points. The CPT total score may range from 0 to 14 points (Spinnler e Tognoni, 1987).
  In the remote assessment the visual stimuli will be displayed on the video using the share screen option. The participant will draw the geometric figures on a blank sheet and then show them to the camera.
Comparison of the remote and face-to-face performance on the oral version of Symbol Digit Modalities Test (SDMT) | Day 1 (t0) and Day 15 (t1)
  The SDMT is used to assess psychomotor speed, which measures processing speed as well as motor speed. Performance is also affected by attention, visual scanning and tracking, and working memory. Individuals are required to use a coded key to match nine abstract symbols paired with numerical digits. The final score is the correct number of substitutions in 90 seconds, and scores range between 0 and 110. Higher scores indicate better performance (Nocentini et al., 2006).

SECONDARY OUTCOMES:
Feasibility and satisfaction degree of people with cognitive disorders and caregivers about the remote neuropsychological assessment | Day 15 (t1)
  The feasibility and satisfaction degree about the remote neuropsychological assessment will be measured by a questionnaire that participants will complete immediately after the second and last evaluation. The questionnaire was developed ad hoc and it consists of 16 six-point Likert Scale questions (from Completely Agree to Completely Disagree) and an open-ended question (feedback or suggestions). A total score will not be calculated. Each item of the survey will be considered individually.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Zucchella, PsyD, Principal Investigator — University Hospital of Verona
Locations (1):
- University Hospital of Verona, Verona, VR, Italy

REFERENCES:
- [Background] Appleman ER, O'Connor MK, Boucher SJ, Rostami R, Sullivan SK, Migliorini R, Kraft M. Teleneuropsychology clinic development and patient satisfaction. Clin Neuropsychol. 2021 May;35(4):819-837. doi: 10.1080/13854046.2020.1871515. Epub 2021 Jan 27. PMID 33504268
- [Background] Wadsworth HE, Dhima K, Womack KB, Hart J Jr, Weiner MF, Hynan LS, Cullum CM. Validity of Teleneuropsychological Assessment in Older Patients with Cognitive Disorders. Arch Clin Neuropsychol. 2018 Dec 1;33(8):1040-1045. doi: 10.1093/arclin/acx140. PMID 29329363
- [Background] Beishon LC, Elliott E, Hietamies TM, Mc Ardle R, O'Mahony A, Elliott AR, Quinn TJ. Diagnostic test accuracy of remote, multidomain cognitive assessment (telephone and video call) for dementia. Cochrane Database Syst Rev. 2022 Apr 8;4(4):CD013724. doi: 10.1002/14651858.CD013724.pub2. PMID 35395108
- [Background] Carotenuto A, Rea R, Traini E, Ricci G, Fasanaro AM, Amenta F. Cognitive Assessment of Patients With Alzheimer's Disease by Telemedicine: Pilot Study. JMIR Ment Health. 2018 May 11;5(2):e31. doi: 10.2196/mental.8097. PMID 29752254
- [Derived] Bressan MM, Musso AM, Bovi T, Bonetti B, Zucchella C. Tele-neuropsychological multidomain assessment in Italian people with cognitive disorders: Reliability and user satisfaction. J Alzheimers Dis. 2025 Jan;103(1):268-281. doi: 10.1177/13872877241300186. Epub 2024 Dec 19. PMID 39702991